CLINICAL TRIAL: NCT01634893
Title: A Phase I Dose-Escalation Trial of Oral Hydroxychloroquine Plus Oral Sorafenib to Treat Patients With Refractory or Relapsed Solid Tumors
Brief Title: Oral Hydroxychloroquine Plus Oral Sorafenib to Treat Patients With Refractory or Relapsed Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRC 11-71; HSC20120203H (Other: UTHSCSA IRB)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Refractory or Relapsed Solid Tumors
Keywords: Refractory or Relapsed Solid Tumors
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib plus Hydroxychloroquine (Experimental): Dose escalation of sorafenib combined with hydroxychloroquine (HCQ) to a maximum of sorafenib 400 mg PO BID plus HCQ 400 mg PO QD.
  Drugs are given on an intermittent schedule of days 1-5/week in a 28-day cycle.
  Sorafenib alone is given in cycle 1, and HCQ is added in cycle 2.
  Interventions: Drug: Sorafenib combined with Hydroxychloroquine

INTERVENTIONS:
Drug: Sorafenib combined with Hydroxychloroquine — dose escalation of sorafenib combined with hydroxychloroquine (HCQ) to a maximum of sorafenib 400 mg PO BID plus HCQ 400 mg PO QD.
  Drugs are given on an intermittent schedule of days 1-5/week in a 28-day cycle.
  Sorafenib alone is given in cycle 1, and HCQ is added in cycle 2.

SUMMARY:
Patients with recurrent, refractory or metastatic solid tumors have a dismal prognosis with few viable treatment options. Hydroxychloroquine (HCQ) is an agent that has been widely used to treat malaria. Because HCQ also inhibits autophagy, a process central to survival of cancer in the face of metabolic stress, including the effects of anti-cancer therapy, it is now in human cancer trials combined with other agents to attempt to boost the efficacy of those agents. Autophagy inhibition improves the activity of sorafenib in hepatocellular carcinoma.

Sorafenib is an oral multi-kinase inhibitor that blocks not only receptor tyrosine kinases such as KIT, VEGFR and PDGFR but also serine/threonine kinases along the RAS/RAF/MEK/ERK pathway.

The investigators propose to treat patients with refractory or relapsed solid tumors with sorafenib, to boost its efficacy while attempting to mitigate its toxicity by combining with HCQ.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Not on immune-modulating drugs, except those used as study drug premedication, unless the principal investigator grants an exception (which exception must be documented in writing)
* Patients with relapsed or refractory solid tumors with no viable treatment options
* Measurable disease within 30 days of study enrollment
* Blood hemoglobin > 8.5 gm/dl within 7 days of study enrollment
* Absolute neutrophil count > 1000/mm3 within 7 days of study enrollment
* Platelet count > 50,000/mm3 within 7 days of study enrollment
* SGOT <10x upper limit of normal within 7 days of study enrollment
* No chemotherapy or radiation therapy in the 14 days prior to initiation of treatment on this study. No other concurrent chemotherapy, surgery or radiation therapy during this protocol except surgery or radiation therapy to control symptoms with concurrence of the principal investigator.
* No contraindication to any study treatment
* No active major medical problems, including untreated or uncontrolled infections
* If of reproductive potential, a negative urine or blood pregnancy test within 3 days of study enrollment, and agreement to use adequate contraception. In relevant subjects, pregnancy testing will continue monthly while on treatment unless the subject is no longer able to become pregnant or there is sufficient justification otherwise
* Not breast feeding
* Life expectancy > 6 months
* ECOG performance status < 2
* Age 18+ years
* No active substance abuse in the prior 6 months
* Not on digoxin or cimetidine

Exclusion Criteria:

* Contraindication or hypersensitivity to any study drug or its components or excipients
* Current pregnancy or breast feeding
* Inability to document adequate contraception if a female of reproductive potential
* Chemotherapy or radiation therapy within the 14 days prior to initiation of study treatment
* Prior treatment with sorafenib. Prior HCQ use is not an exclusion.
* Life expectancy < 6 months
* ECOG performance status > 2
* Symptomatic coronary artery disease (including uncontrolled angina, congestive heart failure, and the like)
* Uncontrolled hypertension (diastolic BP consistently >100 mm Hg or systolic BP consistently >160 mm Hg on a regular basis)
* Uncontrolled, symptomatic cardiac arrhythmia
* Active substance abuse in the prior 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Toxicity evaluated according to the common toxicity criteria for adverse events (AEs) (CTCAEv4.0) | 2 years
  To assess the toxicities of combining sorafenib plus HCQ in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Curiel, MD, MPH, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas, United States